CLINICAL TRIAL: NCT06180252
Title: PET Study of Acetylcholine Esterase Activity in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: MP4-FIN2001
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET with 11C MP4 — Each subject will undergo a PET exam using 11C MP4 as a tracer. This is a specific ligand for the acetyl-choline esterase enzyme already used abroad both in healthy volunteers and in various patient groups.

SUMMARY:
The aim of this study is to understand regional variations in acetylcholine esterase activity in Alzheimer's disease. In this study the aim is to identify by PET the physiological values of the regional activity of acetylcholine esterase using the 11C PM4 tracer and to study by PET and 11C PM4 the brain activity of acetylcholine esterase in a group of patients with Alzheimer's disease, enrolled according to the inclusion and exclusion criteria. The PET data will be correlated with the clinical, neuropsychological and morphological data acquired by MRI and with the clinical-cognitive outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with Alzheimer's disease;
* patients must have undergone an instrumental morphological examination to exclude other neurological pathologies.

Exclusion Criteria:

* positive history of major head trauma;
* clinically active somatic diseases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Alzheimer's disease who are eligible for therapy with acetylcholine esterase inhibitors but not yet undergoing treatment.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-05-12 (Actual); Primary Completion 2008-01-29 (Actual); Study Completion 2008-01-29 (Actual)

PRIMARY OUTCOMES:
PET with 11C MP4 as a tracer to identify acetylcholine esterase values in patients with neurodegenerative diseases. | 4 years
  Development of a new PET method for the in vivo measurement of acetylcholine esterase activity at the cortical level to be used as an indicator of the presence of disease.

IPD SHARING:
Plan to Share IPD: No